CLINICAL TRIAL: NCT07042620
Title: Ultrasound Imaging in Brain Tumour Surgery With the Use of SonoClear® System Mimicking Brain Tissue.
Brief Title: A Study to Test a New Fluid to Improve the Quality of Images Obtained by Using Sound Waves (Ultrasound) During Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SonoClear AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACF-03-02
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Brain Tumor Adult; Low Grade Glioma (LGG), High Grade Glioma (HGG); Glioblastoma
Keywords: Acoustic Coupling Fluid; Ultrasound imaging in brain tumour surgery; brain tumour surgery
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: A prospective, multi-centre single arm study
Masking Description: The following measures have been taken to minimize or avoid bias:
  * Core-lab evaluation of the CNR outcome in a blinded fashion
  * SIR clinical rating of US images by an independent expert panel in a blinded fashion
  Due to the nature of brain surgery and the diversity of the tumours, it is seen as a strength to the trial that the patient can act as its own control even though the images can never be 100% the same in the separate image acquisition. This is especially true for 2D US images, whereas with a 3D US image it is more likely to obtain the same position for sequential image acquisition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound imaging in brain tumour surgery with the use of SonoClear® System mimicking brain tissue. (Experimental): SonoClear(R) System
  Interventions: Device: SonoClear(R) System

INTERVENTIONS:
Device: SonoClear(R) System — The SonoClear(R) System is intended to be used as an acoustic coupling fluid during ultrasound imaging in brain surgery of human beings

SUMMARY:
The objective of this clinical investigation is to assess the safety and performance of the SonoClear® System. Performance will be assessed by analysis of the contrast-to-noise ratio (CNR) and assessment of image quality by using the Surgeon Image Rating (SIR) Scale.

This is a prospective, multi-centre single arm study where the performance of the SonoClear® System relative to routinely used acoustic coupling fluid is investigated by each patient being their own control. Patients with the diagnosis of high-grade glioma (HGG) and low-grade glioma (LGG) at up to 5 sites in Germany will be included. Additionally, safety data are collected at 72 hours, 30 days and 6 months post procedure.

DETAILED DESCRIPTION:
Ultrasound images will be obtained at different timepoints during the operation. First timepoint being after craniotomy (no fluids involved). Second timepoint being when some tumour is left in the bottom of the deeper part of the resection cavity (approximately 80% of tumour removed), and third timepoint being when the surgeon deems resection of the tumour to be completed. At the second and third timepoint ultrasound acquisition will be performed twice at each timepoint. Once with routinely used irrigation fluids (physiologic saline 0.9% / ringer's / lactated ringers' solution) and once with SonoClear® as part of the SonoClear® System

There are two performance related primary endpoints, based on core lab assessments:

1. To assess ultrasound images obtained with SonoClear® as part of the SonoClear® System are less influenced by image artefacts compared to images obtained with standard of care irrigation fluid, by measuring the contrast-to-noise ratio (CNR). The CNR is a measure of the relative noise in the image.
2. To assess ultrasound images obtained with SonoClear® as part of the SonoClear® System compared to images obtained with standard of care irrigation fluids, by using a qualitative assessment, called the Surgeons Image Rating (SIR) scale. A Panel of Experts will assess the quality of the obtained images by answering 3 questions for each image. For SIR a 1-10 numeric rating scale, is used to measure the quality of the image according to three questions to be answered at the three different timepoints during the operation.

This SIR is designed to explore whether SonoClear® as part of the SonoClear® System having shown to provide better quantitative image quality in the CNR analysis, allows surgeons to detect this improved image quality. Eventually this improved image quality should result in better decision-making during surgery about margins of excision and residual tumour resection.

The primary safety event is defined as any core lab determined major Magnetic Resonance Imaging (MRI) finding when post-operative MRI is compared to pre-operative MRI that was found by the Data Monitoring Committee (DMC) to be serious and probably or definitely related to the study device OR any DMC determined serious adverse event that is probably or definitely related to the study device that occurs within 30 days of the procedure. The primary safety hypothesis declared in ACF-03 study is to prove the primary safety event rate is less than 10%. Success is demonstrated by observing 0 of these events out of 37 subjects exposed to SonoClear® ACF, i.e. the event rate is 0% with an upper two-sided 95% confidence limit less than 10%. With an event rate of less than 10% for major neurotoxicity events that are serious and probably or definitely related to the device, the benefit of a clearer image for the neurosurgeon balances the potentially increased risk. This study expands the number of patients to evaluate the safety outcome. The primary safety event rate will be evaluated also in a total group of 60 patients, 45 using SonoClear® ACF and 15 using the SonoClear® System.

ELIGIBILITY:
Key Inclusion Criteria:

* A diffuse malignant glial tumour (high grade (grade III and IV) or low grade (grade I-II)) is suspected from the diagnostic MRI scan
* Pre- or peri-procedural confirmed histopathology of glioma
* ≥18 years of age
* Karnofsky performance status ≥ 70
* Life expectancy of more than 30 days at the time of procedure
* Negative pregnancy test for female subjects of childbearing potential

Key Exclusion Criteria:

* Not able to give consent (e.g., severe cognitive impairment)
* History of brain radiation therapy
* Recent meningitis (within 6 months prior to screening visit)
* Other active infection (within 30 days prior to screening visit)
* Immuno-incompetent patient (e.g., failing immune system due to AIDS)
* Patients taking immune-suppressive medication
* Intended biopsy only (meaning cases not suitable for resection)
* Known hypersensitivity to egg protein
* Known hypersensitivity to soybean or peanut protein
* Known Hypersensitivity to glycerol
* Pregnant or lactating females or females who intend to become pregnant during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Contrast-to-Noise Ratio (CNR) to quantify the reduction in noise | Ultrasound guided brain tumor resection procedure/surgery
  To show that ultrasound images obtained when using the SonoClear(R) System are less influenced by image artefacts compared to images obtained when using routinely used saline solution measuring the contrast-to-noise ratio (CNR) in the images.
Surgeons Image Rating (SIR) to assess the image quality | Ultrasound guided brain tumor resection procedure/surgery
  Quality assessment of the images is done by the core-lab in a blinded manner using the Surgeon Image Rating (SIR) scale, a 1-10 rating scale to score the quality of the image according to 3 questions at different time points during the operation. First timepoint being after craniotomy (no fluids involved). The second time point is when some tumour is left in the bottom of the deeper part of the resection cavity (approximately 80% of tumour removed), and the third time point being when the surgeon deems resection of the tumour to be completed.
Adverse events up to 6 months post procedure | safety data are collected up to 6 months post procedure
  The primary safety hypothesis declared in ACF-03 study is to prove the primary safety event rate is less than 10%. Success is demonstrated by observing 0 of these events out of 37 subjects exposed to SonoClear® ACF, i.e. the event rate is 0% with an upper two-sided 95% confidence limit less than 10%. With an event rate of less than 10% for major neurotoxicity events that are serious and probably or definitely related to the device, the benefit of a clearer image for the neurosurgeon balances the potentially increased risk. This study expands the number of patients to evaluate the safety outcome. The primary safety event rate will be evaluated also in a total group of 60 patients, 45 using SonoClear® ACF and 15 using the SonoClear® System.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Universitätsklinikum Gießen und Marburg GmbH Standort Marburg, Marburg
  - Eberhard Karls Universität Tübingen, Faculty of Medicine, Department of Neurosurgery, Tübingen
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No